CLINICAL TRIAL: NCT06917716
Title: Translation and Validation of a Chinese Version of the Comprehensive Pain Assessment Tool Short Form (COMPAT-SF) in Patients With Chronic Pancreatitis
Brief Title: Translation and Validation of Chinese COMPAT-SF
Acronym: COMPAT-SF-CV
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHEC2025-050
Record Dates: First submitted 2025-03-20; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic Pancreatitis; Pain Assessment; Cross-Cultural Adaptation; Comprehensive Pain Assessment Tool Short Form
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to translate, adapt, and test the reliability of a Chinese version of the Comprehensive Pain Assessment Tool Short Form (COMPAT-SF) for people with chronic pancreatitis.

The study will answer these questions:

* Does the Chinese COMPAT-SF work well to measure pain in people with chronic pancreatitis?
* Is the Chinese COMPAT-SF accurate and reliable over time?

Participants will:

* Complete the Chinese COMPAT-SF questionnaire two times, with a 2-week gap.
* Answer additional pain-related questions using the Brief Pain Inventory (BPI) and the Izbicki Pain Score.
* Participate in a follow-up to check if the questionnaire gives consistent results over time.

This study will help make sure that doctors in China have a useful and reliable tool to measure pain in people with chronic pancreatitis.

DETAILED DESCRIPTION:
This multicenter observational study aims to translate, culturally adapt, and validate the Chinese version of the Comprehensive Pain Assessment Tool Short Form (COMPAT-SF) for individuals with chronic pancreatitis (CP), ensuring it is a reliable and valid pain assessment tool in China.

A total of 356 participants diagnosed with CP will be recruited from Changhai Hospital (Naval Medical University) and Peking Union Medical College Hospital. The study will follow a structured translation process, including forward translation, back translation, expert panel review, and cognitive debriefing to ensure cultural and linguistic appropriateness. Participants will complete the Chinese COMPAT-SF at baseline and again after two weeks to assess test-retest reliability, alongside additional pain assessments using the Brief Pain Inventory (BPI) and Izbicki Pain Score.

Psychometric analysis will evaluate internal consistency (Cronbach's α), test-retest reliability (intraclass correlation coefficient, ICC), construct validity (confirmatory factor analysis, CFA), and criterion validity (correlation with BPI and Izbicki Pain Score). Data will be securely recorded in an electronic database with quality control measures, including predefined range checks, consistency verification, and source data validation against medical records. Standard Operating Procedures (SOPs) will guide participant recruitment, data collection, and statistical analysis, with missing data handled using multiple imputation techniques.

Statistical analyses will include descriptive statistics, Cronbach's α for internal consistency, ICC for reliability, CFA for construct validity, and Pearson correlation to assess criterion validity. This study is expected to provide a scientifically validated, culturally adapted pain assessment tool for chronic pancreatitis, improving clinical evaluation and patient care.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with chronic pancreatitis (CP) according to the Guidelines for the Diagnosis and Treatment of Chronic Pancreatitis in China (2018 edition). Diagnosis can be confirmed by: •Primary diagnostic criteria: (i) Definitive imaging findings, and (ii) Histopathological confirmation. •Secondary diagnostic criteria: (i) Recurrent upper abdominal pain, (ii) Abnormal serum amylase levels, (iii) Pancreatic exocrine insufficiency, (iv) Pancreatic endocrine insufficiency, (v) Pathogenic gene mutations, and (vi) History of heavy alcohol consumption. •Diagnosis is confirmed if at least one primary criterion or two secondary criteria are met.
* 2. Experience of pancreatic pain in the past 12 months

Exclusion Criteria:

* Under 18 years of age.
* No pancreatic-related pain.
* Diagnosed with pancreatic cancer or other tumors.
* Presence of communication or reading impairments.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit individuals diagnosed with chronic pancreatitis (CP) experiencing pancreatic pain from Changhai Hospital and Peking Union Medical College Hospital. Eligible participants are those who meet the diagnostic criteria outlined in the Guidelines for the Diagnosis and Treatment of Chronic Pancreatitis in China (2018 edition) and have experienced pancreatic pain in the past 12 months. The study will be conducted between March 2025 and June 2026, enrolling participants during their hospital visits.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency of COMPAT-SF-CV | Baseline
  Internal consistency will be evaluated using Cronbach's alpha for each domain and the total score of the Chinese version of the Comprehensive Pain Assessment Tool Short Form (COMPAT-SF-CV).
Test-Retest Reliability of COMPAT-SF-CV | Baseline and 2-week follow-up
  Test-retest reliability will be assessed using intraclass correlation coefficient (ICC) between baseline and 2-week follow-up responses on COMPAT-SF-CV.
Construct Validity of COMPAT-SF-CV | Baseline
  Construct validity will be examined through confirmatory factor analysis (CFA) to assess the underlying factor structure of COMPAT-SF-CV.
Criterion Validity of COMPAT-SF-CV | Baseline
  Criterion validity will be assessed by calculating correlations between COMPAT-SF-CV scores and established measures of pain severity, including the Brief Pain Inventory (BPI) and Izbicki pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No